CLINICAL TRIAL: NCT05842824
Title: An Observational Study of Patients With Autoimmune Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-AUTOIMMUNE
Record Dates: First submitted 2023-03-09; First posted 2023-05-06 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-04

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease Cohort: Observational
- Engaged Cohort: Observational

SUMMARY:
TARGET-AUTOIMMUNE is an observational research study to conduct a comprehensive review of outcomes for patients with autoimmune and related diseases. .

ELIGIBILITY:
Disease Cohort

Inclusion Criteria:

- Adult patients at the time of enrollment with a diagnosis autoimmune disease by select ICD-10 codes in the EHR interface

Exclusion Criteria:

* Death
* Manual removal (sponsor or site request)
* No EHR interface encounter > 3 years

Engaged Cohort

Inclusion Criteria:

* Adult patients diagnosed and managed for these conditions invited to participate
* Ability to provide written informed consent

Exclusion Criteria:

* Patient expressed desire to withdraw consent to complete PROs
* Failure to complete PROs within 24 weeks of initial invitation
* Greater than 24 months lapse of survey completion after baseline surveys completed
* Additionally, the criteria detailed for Disease Cohort apply to the Engaged Cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adults who are being managed for autoimmune disease
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2038-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
To characterize the natural history of disease in patients with autoimmune disease of various etiologies. | 15 Years
To assess safety and effectiveness of autoimmune disease treatments and treatments for complications of any related conditions | 20 Years

SECONDARY OUTCOMES:
To evaluate provider management practices in the treatment of patients with autoimmune diseases | 15 Years
  Health care provider type, clinic setting, reason for initiating/not initiating/adjusting dosing of treatments, reason for discontinuing/switching treatments, and monitoring outcomes on and off treatment, will be captured as available in the provided EHR and/or through linked data. Disease-specific quality measures will be selected and evaluated.
To evaluate longitudinal and patient reported outcomes in patients with autoimmune diseases | 15 Years
  Longitudinal clinical outcomes and disease progression will be assessed. Self-reported patient health measures collect information directly from patients to measure physical, mental, and social health. These measures can help clinicians better understand how the disease state and/or various treatments affect what patients are able to do and the symptoms they experience beyond what is typically derived and reported in the EHR as part of traditional clinical evaluations. The information can also be used to help patients make informed decisions about their healthcare and treatment options.
To select and evaluate quality of care measures for patients with autoimmune diseases | 15 Years
  1. Identify and select best practices in care of patients with autoimmune diseases
  2. Develop a technology infrastructure to evaluate quality measures to support clinicians.

IPD SHARING:
Plan to Share IPD: Undecided